CLINICAL TRIAL: NCT04012970
Title: The Investigation of Muscle Stiffness, Tone and Elasticity After a Spinal Mobilisation Intervention in People With Lower Back Pain
Brief Title: Investigating the Effects of a Spinal Mobilisation Intervention in People With Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edinburgh Napier University (Other)
Collaborators: Scottish Hospital Endowments Research Trust (Other); Pacla Medical Limited (Industry)
Responsible Party: Principal Investigator, Rebecca Hamilton, Principal Investigator, PhD student, Edinburgh Napier University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PILOT_LBP_1
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Lower Back Pain
Keywords: lower back pain; myometer; muscle stiffness; spinal mobilisations
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Cross-over study design, within-subject repeated measures (intervention versus no intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Intervention then control (Experimental): Intervention (30 minutes spinal mobilisations) received in first session, then control (30 minutes lying still) received in second session.
  Interventions: Other: Manual spinal mobilisations
- B - Control then intervention (Experimental): Control (30 minutes lying still) received in first session, then intervention (30 minutes spinal mobilisations) received in second session.
  Interventions: Other: Manual spinal mobilisations

INTERVENTIONS:
Other: Manual spinal mobilisations

SUMMARY:
The objective of the study is to measure and analyse the effect of a spinal mobilisation intervention on muscle tissue quality in people with lower back pain. The mobilisation intervention will be compared to a control with participants taking part in both conditions for a factorial, within-subject repeated measures study. The study will analyse lumbar muscle response to the manual intervention and analyse the potential influence of anthropometric measures of participants. The study hypothesises a decrease in lumbar stiffness post the intervention, compared to the control session.

DETAILED DESCRIPTION:
Various types of spinal manual therapies have been common practice for many years, particularly for treatment of lower back pain. Spinal mobilisation is a specific technique within spinal physiotherapy, often used as a treatment for lower back pain. This is despite limited objective evidence of the effect on muscle tissue quality.

The objective of this study is to measure and analyse the acute effect of a spinal mobilisation intervention on muscle tissue quality in people with lower back pain. The intervention consists of the mobilisation of the lumbar spine for 30 minutes, at a specific rate and pressure. This will be performed by a chartered physiotherapist. This will be tested with 40 participants with lower back pain. This was the recommended sample size given by G Power for a medium effect size, a power of 0.95 and alpha level of 0.05.

Participants will take part in an intervention and a control condition. Lumbar muscle response will be measured for stiffness, tone and elasticity immediately before and after the intervention and the control. The control session consists of lying still for the 30 minutes. Results for both sessions will then be compared. A myometer (MyotonPRO) will be used to assess the change in lumbar muscle objectively. This is a non-invasive, handheld device with many reliability studies on its functionality. Analysis will consider the degree of muscle response with individual covariates involved. This includes gender, height, weight, waist circumference, BMI and level of back pain (discerned by score on Oswestry Disability Index).

The results will compared in 2-way repeated measures, within participant ANOVA for significant differences between conditions and time. Anthropometric measures will be analysed in separate ANOCOVAs to determine any significant factors contributing to level of change.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from lower back pain (region between 12th rib and gluteal folds), acute or chronic.

Exclusion Criteria:

Respond positively to any absolute contraindications for spinal therapy, including:

* segment instability
* infectious disease
* osteomyelitis
* bone tumours
* neurological deficit
* upper motor neuron lesion
* spinal cord damage
* cervical arterial dysfunction

Respond positively to relative contra-indications, excluded based on severity, including:

* osteoporosis
* spinal instability
* rheumatoid arthritis
* inflammatory disease
* active history of cancer
* hypermobile syndrome
* segment hypermobility
* cardiovascular disease
* cervical anomalies
* nerve root disorder
* spinal surgery
* respiratory problems
* thrombosis
* open wounds
* local infection
* fractures or dislocations

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Brown, Study Director — Director of PhD Studies
Locations (1):
- Edinburgh Napier University, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant data sets that underlie the results for publication will be shared on a raw data set. This includes the muscle quality data, back pain result, and anthropometric data.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be entered when the study is completed and remain until 1 year post publication of summary data.
Access Criteria: The anonymised participant data underlying the summary data published, will be shared on the Edinburgh Napier University Repository with submission of PhD thesis.

RESULTS

PARTICIPANT FLOW:
Groups:
- A - Intervention Then Control: Intervention (30 minutes spinal mobilisations) received in first session, control (30 minutes lying still) received in second session.
Period: Intervention Session, 30 Minutes
Arm/Group | A - Intervention Then Control | B - Control Then Intervention
Started | 26 | 14
Completed | 26 | 14
Not Completed | 0 | 0
Period: Control Session, 30 Minutes
Arm/Group | A - Intervention Then Control | B - Control Then Intervention
Started | 26 | 14
Completed | 26 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Intervention Then Control | B - Control Then Intervention | Total
Number analyzed (Participants) | 26 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.73 (12.99) | 28 (6.92) | 31.075 (11.373)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 13 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Intervention Erector Spinae Stiffness Change
Description: Stiffness values measured before and after 30 minute spinal mobilisation intervention. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle stiffness immediately after the 30 minute spinal mobilisation intervention.
Measure: Mean (Standard Error); unit: Newton metres (Nm)
Groups:
- Intervention: Group A and Group B results for stiffness change due to the spinal mobilisation intervention.
Arm/Group | Intervention
Number analyzed (Participants) | 40
Newton metres (Nm) | -10.959 (4.132)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p < 0.05, ANOVA; 2-way, repeated measures
Statistical Analysis 2: Comparison: Intervention; Stiffness change ran with covariates (baseline stiffness, BMI, ODI, waist circumference, height and gender); Test type: Superiority; p < 0.01, ANCOVA

2. Primary Outcome: Control Erector Spinae Stiffness Change.
Description: Stiffness values measured before and after 30 minute control lying still. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle stiffness immediately after the 30 minute control session (lying still).
Measure: Mean (Standard Error); unit: Newton metres (Nm)
Groups:
- Control: Group A and Group B results for stiffness change due to the control session.
Arm/Group | Control
Number analyzed (Participants) | 40
Newton metres (Nm) | 12.192 (4.023)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p < 0.01, ANOVA; 2-way, repeated measures
Statistical Analysis 2: Comparison: Control; Stiffness change ran with covariates (baseline stiffness, BMI, ODI, waist circumference, height and gender); Test type: Superiority; p < 0.01, ANCOVA

3. Secondary Outcome: Intervention Erector Spinae Tone Change
Description: Tone values measured before and after 30 minute spinal mobilisation intervention. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle tone immediately after the 30 minute spinal mobilisation intervention.
Measure: Mean (Standard Error); unit: Hertz (Hz)
Groups:
- Intervention: Group A and Group B results for tone change due to the spinal mobilisation intervention.
Arm/Group | Intervention
Number analyzed (Participants) | 40
Hertz (Hz) | -0.317 (0.088)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p < 0.01, ANOVA; 2-way, repeated measures
Statistical Analysis 2: Comparison: Intervention; Tone change ran with covariates (baseline stiffness, BMI, ODI, waist circumference, height and gender); Test type: Superiority; p < 0.05, ANCOVA

4. Secondary Outcome: Control Erector Spinae Tone Change
Description: Tone values measured before and after 30 minute control lying still. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle tone immediately after the 30 minute control session (lying still).
Measure: Mean (Standard Error); unit: Hertz (Hz)
Groups:
- Control: Group A and Group B results for tone change due to the control session.
Arm/Group | Control
Number analyzed (Participants) | 40
Hertz (Hz) | 0.29 (0.1)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p < 0.01, ANOVA; 2-way, repeated measures
Statistical Analysis 2: Comparison: Control; Tone change ran with covariates (baseline stiffness, BMI, ODI, waist circumference, height and gender); Test type: Superiority; p < 0.05, ANCOVA

5. Secondary Outcome: Intervention Erector Spinae Elasticity Change
Description: Elasticity values measured before and after 30 minute spinal mobilisation intervention. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. The device records the logarithmic decrement of the tissue by recording the dissipation of the mechanical energy of the tissue when it recovers shape after deformation. Elasticity is then inversely proportional to the decrement, so a higher decrement value equates to a higher dissipation of mechanical energy and a lower elasticity value. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle elasticity immediately after the 30 minute spinal mobilisation intervention.
Measure: Mean (Standard Error); unit: Logarithmic decrement
Groups:
- Intervention: Group A and Group B results for elasticity change due to the spinal mobilisation intervention.
Arm/Group | Intervention
Number analyzed (Participants) | 40
Logarithmic decrement | 0.068 (0.02)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p < 0.01, ANOVA; 2-way, repeated measures

6. Secondary Outcome: Control Erector Spinae Elasticity Change
Description: Elasticity values measured before and after 30 minute control lying still. Location of muscle assessed by palpation by asking participant to contract lower back muscles and marking the central belly of the muscle. Myometer measurements recorded using handheld device MyotonPRO held over marked area. The device records the logarithmic decrement of the tissue by recording the dissipation of the mechanical energy of the tissue when it recovers shape after deformation. Elasticity is then inversely proportional to the decrement, so a higher decrement value equates to a higher dissipation of mechanical energy and a lower elasticity value. Recorded 3 times and mean value used for analysis.
Time Frame: Change in muscle elasticity immediately after the 30 minute control session (lying still).
Measure: Mean (Standard Error); unit: Logarithmic decrement
Groups:
- Control: Group A and Group B results for elasticity change due to the control session.
Arm/Group | Control
Number analyzed (Participants) | 40
Logarithmic decrement | 0.05 (0.012)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p < 0.001, ANOVA; 2-way, repeated measures

ADVERSE EVENTS:
Time Frame: 1 hour testing time from baseline to post intervention, and 1 hour testing time on separate occasion 1 week apart from baseline to post control.
Description: The intervention consisted of a gentle grade manual therapy, with no serious side effect risk.
Groups:
- Group A - Intervention: Group A received the 30 minutes spinal mobilisations intervention in the first session.
- Group A - Control: Group A received the control (30 minutes lying still) in the second session.
- Group B - Intervention: Group B received the control (30 minutes lying still) in the second session.
  .
- Group B - Control: Group B received the 30 minutes spinal mobilisations intervention in the first session.
Arm/Group | Group A - Intervention | Group A - Control | Group B - Intervention | Group B - Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Variation in level of lower back pain participants was low. Physical activity was not controlled and could be a factor in baseline muscle measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT04012970/Prot_SAP_000.pdf